CLINICAL TRIAL: NCT01985243
Title: Building Capacity for Sustainable Livelihoods and Health Through Public-private Linkages in Agriculture and Health Systems
Brief Title: Building Capacity for Sustainable Livelihoods and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Foreign Affairs, Trade and Development, Canada (Other); World Vision (Other)
Responsible Party: Principal Investigator, Grace S. Marquis, Associate Professor, Canadian Research Chair in Social and Environmental Aspects of Nutrition, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S065653
Record Dates: First submitted 2013-10-27; First posted 2013-11-15 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Malnutrition; Anemia
Keywords: Dietary diversity; Infant and young child; Adolescents; Anemia; Rural health
MeSH Terms: conditions — Malnutrition; Anemia | interventions — Nutritional Status; Agriculture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nutrition and agriculture (Experimental): Intervention arm with integrated nutrition and agriculture education, skill building, and animal husbandry promotion
  Interventions: Behavioral: Nutrition and agriculture
- Iron-rich food & business literacy (Experimental): Integrated business literacy and food supplementation program to promote school retention among female adolescents
  Interventions: Behavioral: Iron-rich food & business literacy
- IYC Comparison (No Intervention): Comparison group of infants and young children for the nutrition-agriculture intervention
- Adolescent comparison (No Intervention): Comparison group for the adolescent business-food supplement intervention

INTERVENTIONS:
Behavioral: Nutrition and agriculture — The intervention includes two components: (1) nutrition education on infant and young child nutrition, and (2) agriculture and small animal husbandry intervention to increase women's income and the accessibility of animal source foods for infants and young children.
  Arms: Nutrition and agriculture
Behavioral: Iron-rich food & business literacy — The intervention includes two components: (1) a behavioural change intervention to improve school meals and increase the available iron in adolescents' diets, (2) savings & business literacy program for young female adolescents to encourage them to stay in school.
  Arms: Iron-rich food & business literacy

SUMMARY:
Despite recent economic growth in Ghana, the prevalence of childhood malnutrition remains high. Wasting prevalence affected 29% among 6- to 8-months-old infants in 2008. Poor nutrition contributes to about one-third of child mortality, diminishes cognitive development, and is a major determinant of maternal mortality. The specific objectives of the 5-year project are to: (1) enhance human capacity of government, civil, and private institutions through improvement of knowledge and skills of personnel in agriculture, nutrition and health, entrepreneurship, and pedagogy; (2) identify information needs of local institutions that are not presently met and develop a representative and sustainable longitudinal data system to support evidence-based decision-making in programs; (3) increase vulnerable households' access to quality services in agriculture/fisheries, nutrition and health, and finance; (4) implement integrated intervention activities to improve infant and young child and adolescent nutrition outcomes; and (5) examine differential benefits of the interventions for diverse vulnerable populations. The project comprises two major activities: part I - the creation of a longitudinal data system to support evidence-based decision-making in programs, and part II - the implementation of intervention activities to improve nutrition outcomes.

The survey will include demographic, socioeconomic, health, diet, and nutritional status information collected annually from a representative same of 1500 households with infants (0-12 mo) and 1500 households with adolescents (9-12 y). The data will be analyzed and presented rapidly each year to district program and policy leaders to assist them in developing their activity plans for the following year.

DETAILED DESCRIPTION:
This study will develop a district-level intervention package that builds capacity of local institutions to improve economic well-being, food security, health and social and cognitive development of populations living in rural Upper Manya Krobo District (UMKD) of Ghana. The UMKD Geographic Information Systems Registry estimates a rural population of 74,290 in 190 communities.

Selection process:

1. Of those UMKD communities that are accessible, 136 communities will be randomly selected.
2. All households with infants 0-12 mo of age in a village will be invited to be enrolled. We will continue to enroll households until we reach our sample size of 1500 households. If necessary, we will expand our number of sampled communities.
3. All households with adolescents 10-15 y of age in a village, who are not part of the infant cohort, will be invited to be enrolled. We will continue to enroll households until we reach our sample size of 1500 households.

Enrollment The survey will be carried out over one day for each community. The field staff will briefly explain the purpose and study activity to the caregiver (parent or legal guardian who is responsible for the child) of the target child. If the caregiver is interested in participating, they will be given the consent form to read, or if illiterate, the consent form will be read to them. They will be given time to ask questions and decide if they wish to participate. For those who consent, they will sign the consent form or provide their finger print as proof of consent. Adolescents will be asked to provide assent. Only once consent (and assent for adolescents) is obtained, will the field staff begin the survey.

Data collection

The annual survey will consist of questions (drafts are attached) on:

1. the household demographics, socioeconomic status, agricultural production, government services use,
2. mother's caregiving practices, microcredit use, business activities, physical and mental health, anthropometry (weight, height), iron status
3. infant's diet, anthropometry (weight, height, circumference), iron status
4. adolescent's diet, anthropometry (weight, height, circumference), iron status, educational activities, finance knowledge

The survey will be administered in the home with the child's caregiver, in a private location. THe adolescent will be interviewed privately unless the mother requests to be present. It is expected to be about 60-90 minutes in length. All data will be recorded solely with the study identification number. The participant's name and home address will be kept secure and separately.

THe interventions will take place with a subgroup of those participating in the annual survey. Our two main integrated interventions target critical periods of the life course when gender inequalities can have important effects on the short-term and long-term health of both men and women. Our first intervention which will begin in January 2014 will offer intensive nutrition, health, and agricultural training, along with provision of home gardens and small animal husbandry to about 302 of our households with at least one child under the age of 1 y. As these will be household-level interventions, both men and women and male and female infants (and older siblings) living in these households will benefit from this intervention. We will assess the extent to which women retain decision-making authority about the allocation of these agricultural resources and whether they benefit their children's health and nutrition, using our primary indicators of child diet and nutritional status.

Our second integrated intervention will focus on reducing anemia among female school-aged children. The intervention will start after the baseline with the beginning of the school year, September 2014. These interventions will benefit both girls and boys as boys also suffer from high rates of anaemia in this district and both sexes continue to have a high burden of parasitic infections. In addition, since older girls (starting in primary grade 4) are less likely to stay in school and, hence, are disadvantaged with respect to their access to these programs, we plan to implement a savings account intervention for girls who successfully complete primary grade 5. The amount of the savings account will be relatively small (e.g., to cover school uniforms) but along with opening these savings accounts girls will gain financial literacy and learn the importance of savings accounts and budgets. Increasing girls' education is one of the most effective ways to decrease child mortality. According to a recent study, about half of the decline in child mortality in developing countries since 1979 can be attributed to women's increased education. Moreover, since our integrated intervention will include means to improve iron status of the girls, , we expect to significantly lower rates of preconception rates of anaemia among these girls. This intervention will help meet one of the key recommendations of The Lancet Maternal and Child Nutrition Series, which notes that "A clear need exists to introduce promising evidence-based interventions in the preconception period and in adolescents in countries with a high burden of undernutrition and young age at first pregnancies" .

ELIGIBILITY:
Inclusion Criteria:

* household with infant < 12 mo or adolescent 10-15 y
* Living in selected communities of Upper Manya Krobo District (Ghana)

Exclusion Criteria:

* infant or adolescent has medical condition that limits dietary intakes or growth

Ages: 1 Day to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3390 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
Dietary diversity | At enrollment and every 12 months for 5 years
  Dietary diversity of infants and young children, based on the World Health Organization's 7 food group list. This will be assessed at enrollment (which 0-11.9 mo of age) and then every 12 months for 5 years.
Anemia prevalence | at enrollment and every 12 months for 4 years
  Anemia prevalence in adolescent girls will be assessed at enrollment and every 12 months for 4 years

SECONDARY OUTCOMES:
Wasting prevalence | at enrollment and every 12 months for 5 years
  Weight-for-height of infants and young children will be assessed at at enrollment and every 12 months for 5 years

OTHER OUTCOMES:
Women's income | at enrollment and every 12 months for 5 years
  Income-generation of child bearing-aged women will be assessed at enrollment and every 12 months for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Marquis, PhD, Principal Investigator — McGill University; Esi K Colecraft, PhD, Principal Investigator — University of Ghana; Bridgett Aidams, PhD, Principal Investigator — World Vision
Locations (3):
- Canada (2):
  - World Vision, Toronto, Ontario
  - McGill University, Montreal, Quebec
- University of Ghana, Legon, Ghana

REFERENCES:
- [Derived] Goh YE, Marquis GS, Colecraft EK, Aryeetey R. Participating in a Nutrition-Sensitive Agriculture Intervention Is Not Associated with Less Maternal Time for Care in a Rural Ghanaian District. Curr Dev Nutr. 2022 Sep 29;6(10):nzac145. doi: 10.1093/cdn/nzac145. eCollection 2022 Oct. PMID 36475016
- [Derived] Dallmann D, Marquis GS, Colecraft EK, Kanlisi R, Aidam BA. Maternal Participation Level in a Nutrition-Sensitive Agriculture Intervention Matters for Child Diet and Growth Outcomes in Rural Ghana. Curr Dev Nutr. 2022 Feb 1;6(3):nzac017. doi: 10.1093/cdn/nzac017. eCollection 2022 Mar. PMID 35295712